CLINICAL TRIAL: NCT03608553
Title: A Study to Evaluate the Safety and Feasibility of Temporary Blood Brain Barrier Disruption (BBBD) Using Exablate MR Guided Focused Ultrasound in Patients With Parkinson's Disease Dementia
Brief Title: A Study to Evaluate Temporary Blood Brain Barrier Disruption in Patients With Parkinson's Disease Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD008
Record Dates: First submitted 2018-03-01; First posted 2018-08-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Parkinsons Disease With Dementia
Keywords: MRgFUS; BBB; Blood Brain Barrier Disruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ExAblate (Experimental): ExAblate MR Guided Focused Ultrasound
  Interventions: Device: MR Guided Focused Ultrasound

INTERVENTIONS:
Device: MR Guided Focused Ultrasound — Blood Brain Barrier Disruption using FUS
  Other Names: ExAblate

SUMMARY:
The goal of this prospective, non-randomized, single-arm, feasibility study is to develop data to evaluate the safety and initial efficacy of this treatment (temporary disruption of the BBB) using this ExAblate Model 4000 Type 2 System in patients with mild to moderate Parkinson´s Disease Dementia

DETAILED DESCRIPTION:
This study is a prospective, single-arm, non-randomized, safety and feasibility trial of focal BBB disruption using the ExAblate® Model 4000 Type 2 (220 kHz) system with Luminity® ultrasound contrast in 10 patients with mild to moderate Parkinson's Disease Dementia. Patients, together with their caregivers, will be approached after their identification by a team of neurosurgeons and neurologists who specialize in the management of cognitive disorders and functional neurosurgery. The study will be discussed with them, and all patients, or their legal representatives will provide informed consent to participate in the study.

This first in human trial will be divided into two stages. In the first stage, patients will undergo small volume BBB disruption, establishing the minimum required sonication parameters to open the BBB, as evidenced by gadolinium enhancement on T1-weighted MRI. Stage I is defined as a discrete region of approximately 9 mm x 9 mm area in the right parietooccipitotemporal cortex. Multiple sonications will be performed starting at low energy and ramping up until the BBB is observed to open.

The subjects will then be removed from the ExAblate® Neuro device and followed for safety for 2 weeks. If the subject experienced BBB disruption without any serious adverse effects (such as brain edema), then the subject may proceed to Stage II where a larger volume (2.5-3.0 cm) will be targeted. Subjects will be followed for an additional 2 weeks for safety and preliminary effectiveness.

The staged approach will allow determination of:

1. Safety of BBB disruption
2. Feasibility of disruption the BBB
3. Reversibility of BBB disruption
4. Reproducibility of BBB disruption

ELIGIBILITY:
Primary Inclusion Criteria:

1. Parkinson´s Disease, according to the UK Parkinson´s Disease Society Brain Bank (Gelb et al. 1999)
2. Parkinson´s Disease patients diagnosed with mild-moderate dementia according to the Movement Disorders Criteria (Emre et al. 2007)
3. Able and willing to give informed consent, or has delegated this to a substitute decision maker.
4. Mini Mental State Exam (MMSE) scores ≥16 (able to complete a Neuropsychological evaluation)
5. Geriatric Depression Scale (GDS) score of ≤ 20
6. Age: 60-80 years
7. Able to attend all study visits (i.e., life expectancy of 1 year).

Primary Exclusion Criteria:

1. Clips or other metallic implanted objects in the skull or the brain, except shunts
2. Significant cardiac disease or unstable hemodynamic status
3. Uncontrolled hypertension (systolic > 150 and diastolic BP > 100 on medication)
4. Medications known to increase risk of hemorrhage, (e.g.: patients should be off of ASA for at least 7 days prior to treatment) or anticoagulants
5. History of a bleeding disorder
6. Significant depression and at potential risk of suicide
7. Known sensitivity/allergy to gadolinium
8. Any contraindications to MRI scanning
9. History of seizure disorder or epilepsy
10. History of drug or alcohol use disorder who may be at higher risk for seizure, infection, or poor executive functioning
11. Chronic breathing disorders

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related Adverse Events as assessed by patient examination and MR imaging | Treatment through Day 14 after Second Treatment
  Adverse events will be categorized according to severity, relationship to surgical procedure, and relationship to ExAblate device.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Obeso, MD, PhD, Principal Investigator — Director of CINAC
Locations (1):
- HM Hospitales Puerta del Sur - CINAC, Móstoles, Madrid, Spain

REFERENCES:
- [Derived] Pineda-Pardo JA, Gasca-Salas C, Fernandez-Rodriguez B, Rodriguez-Rojas R, Del Alamo M, Obeso I, Hernandez-Fernandez F, Trompeta C, Martinez-Fernandez R, Matarazzo M, Mata-Marin D, Guida P, Duque A, Albillo D, Plaza de Las Heras I, Montero JI, Foffani G, Toltsis G, Rachmilevitch I, Blesa J, Obeso JA. Striatal Blood-Brain Barrier Opening in Parkinson's Disease Dementia: A Pilot Exploratory Study. Mov Disord. 2022 Oct;37(10):2057-2065. doi: 10.1002/mds.29134. Epub 2022 Jun 28. PMID 35765711
- [Derived] Gasca-Salas C, Fernandez-Rodriguez B, Pineda-Pardo JA, Rodriguez-Rojas R, Obeso I, Hernandez-Fernandez F, Del Alamo M, Mata D, Guida P, Ordas-Bandera C, Montero-Roblas JI, Martinez-Fernandez R, Foffani G, Rachmilevitch I, Obeso JA. Blood-brain barrier opening with focused ultrasound in Parkinson's disease dementia. Nat Commun. 2021 Feb 3;12(1):779. doi: 10.1038/s41467-021-21022-9. PMID 33536430